CLINICAL TRIAL: NCT04797819
Title: Elevated Serum Soluble ST2 Level is Associated With Increased Plaque Vulnerability in Patients With Non-ST Elevation Acute Coronary Syndrome
Brief Title: Serum Soluble ST2 and Plaque Vulnerability in Patients With Acute Coronary Syndrome
Status: Completed | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: sST2 and plaque vulnerability
Record Dates: First submitted 2021-03-12; First posted 2021-03-15 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Acute Coronary Syndrome
Keywords: soluble ST2; plaque vulnerability
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Serum sST2 level < 14.5 ng/mL
  Interventions: Diagnostic Test: Coronary plaque components
- 14.5 ng/mL ≤ Serum sST2 level < 20.5 ng/mL
  Interventions: Diagnostic Test: Coronary plaque components
- 20.5 ng/mL ≤ Serum sST2 level < 25.9 ng/mL
  Interventions: Diagnostic Test: Coronary plaque components
- Serum sST2 level ≥ 25.9 ng/mL
  Interventions: Diagnostic Test: Coronary plaque components

INTERVENTIONS:
Diagnostic Test: Coronary plaque components — Coronary plaque components were detected by CCTA method

SUMMARY:
This study aimed to assess the association between serum sST2 level and plaque vulnerability in ACS patients. It is hypothesized that serum sST2 level may be related to plaque components and closely associated with plaque vulnerability.

DETAILED DESCRIPTION:
Serum soluble suppression of tumorigenicity-2 (sST2) has emerged as a novel biomarker of atherosclerotic disease. This study aimed to investigate whether elevated serum sST2 level is related to coronary plaque components detected on coronary computed tomography angiography (CCTA) and plaque vulnerability in non-ST elevation acute coronary syndromes (ACS) patients. 167 lesions in 120 non-ST elevation ACS patients were prospectively enrolled and evaluated by CCTA in this study. Blood were taken from antecubital vein during patient's hospitalization for angiography. Serum sST2 level was measured by commerical ELISA kits (Presage ST2 Assay Kit, Critical Diagnostics). CCTA were performed using a 320-slice CT scanner (Aquilion ONE, Toshiba Medical Systems, Otawara, Japan). Coronary plaque components were analyzed cross each of the lesions using commercialized software package (QAngio CT, Medis, The Netherlands).

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of non-ST-elevation ACS

   1. Non-ST-elevation myocardial infarction
   2. Unstable angina
2. Age from 18 to 75 years
3. Underwent CCTA

Exclusion Criteria:

1. Patients needed an immediate (< 2 h) or early invasive strategy (< 24 h) according to guidelines:

   1. Haemodynamic instability
   2. Cardiogenic shock
   3. Life-threatening arrhythmias or cardiac arrest
   4. Mechanical complication
   5. Acute heart failure
   6. Dynamic ST or T wave changes
   7. GRACE score > 140
2. Patients with previous history of:

   1. Coronary artery bypass graft surgery or percutaneous coronary intervention (PCI)
   2. Immune system disorder
   3. Tumor
   4. Acute/chronic infection
   5. Statin use within 3 months
   6. Atrial fibrillation
   7. End-stage renal failure
   8. Iodine-containing contrast allergy
3. Patients with no significant (≥ 50%) stenosis on major epicardial vessels after CCTA performance
4. Patients refused subsequent angiography after CCTA performance
5. Patients with total obstruction on major epicardial vessel
6. Patients with insufficient image quality for QAngioCT analysis

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Between January 2019 and December 2019, a total of 120 patients with 167 lesions were included in our study for final analysis.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Distribution of plaque components by QAngioCT | Procedure (Coronary CTA )
  Hounsfield unit (HU) -30 to 75 for necrotic core, HU 76-130 for fibrous fatty, HU 131-350 for fibrous tissue, and HU over 351 for dense calcium.

CONTACTS AND LOCATIONS:
Overall Officials: Song Ding, Principal Investigator — RenJi Hospital
Locations (1):
- Cardiology, Ren Ji Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Luo G, Qian Y, Sheng X, Sun J, Wu Z, Liao F, Feng Q, Yin Y, Ding S, Pu J. Elevated Serum Levels of Soluble ST2 Are Associated With Plaque Vulnerability in Patients With Non-ST-Elevation Acute Coronary Syndrome. Front Cardiovasc Med. 2021 Jul 22;8:688522. doi: 10.3389/fcvm.2021.688522. eCollection 2021. PMID 34368249